CLINICAL TRIAL: NCT03041740
Title: A Pilot Study to Evaluate the Safety of Perflurooctylbromide (PFOB) Partial Liquid Ventilation (PLV) for Up to 10 Days in Neonates With Severe Bronchopulmonary Dysplasia (BPD)
Brief Title: Fluid Filled Lung Oxygenation Assistance Trial
Acronym: FFLOAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Auto Dealers Caring for Kids Foundation (Other)
Responsible Party: Principal Investigator, William Fox, Attending Physician, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-008686
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — perflubron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Usual Care (Control) Group (No Intervention): Control subjects will be treated as per standard of care for preterm infants with BPD.
- Perfluorooctylbromide (PFOB) Group (Active Comparator): Subjects in the PFOB group will be administered an initial PFOB treatment dose of 2.5 mL/kg and up to a total intra-pulmonary volume of 25 mL/kg for up to 10 days.
  Interventions: Drug: Perfluorooctyl Bromide

INTERVENTIONS:
Drug: Perfluorooctyl Bromide — Subjects in the PFOB group will receive PFOB partial liquid ventilation instilled via side port of endotracheal tube (2.5 mL/kg/day) across 10 treatment days.
  Other Names: Perflubron
  Arms: Perfluorooctylbromide (PFOB) Group

SUMMARY:
The primary study objective is to assess the safety and feasibility of perfluorooctylbromide (PFOB) partial liquid ventilation (PLV) in infants with severe Bronchopulmonary Dysplasia (BPD).

DETAILED DESCRIPTION:
The primary study objective is to assess the safety and feasibility of perfluorooctylbromide (PFOB) partial liquid ventilation for up to ten days in infants with severe BPD as evaluated by: (1) no sustained oxygen desaturations (SpO2 ≤ 80%) for greater than ten minutes without response to increased oxygen therapy, (2) no persistent hypotension without response to volume expansion and/or inotropic therapy, (3) no major mucus plugging events (defined as events that are unresolved after two bronchoscopes), (4) no pneumothoraces or pleural effusion with PFOB, (5) and no evidence of increased carbon dioxide (CO2) retention, renal insufficiency, hyperkalemia, or metabolic acidosis.

ELIGIBILITY:
Inclusion Criteria

1. Neonates with severe BPD as defined by 36 weeks post conception age and require positive pressure ventilation
2. Infants born at less than 32 weeks post conception age
3. Subjects may be up to 6 months corrected age
4. On conventional mechanical ventilation for chronic lung disease for at least two days prior to enrollment
5. On conventional mechanical ventilation at the time of enrollment and anticipated to continue for 14 days
6. Off systemic steroids for lung disease for 72 hours (3 days) prior to T=0
7. Hemoglobin value ≥8 g/dL: if less than 8 g/dL, transfusion is permitted. Clinical blood transfusion should be administered prior to enrollment.
8. Parental/guardian permission (informed consent)

Exclusion Criteria

1. Mechanical ventilation for acute disease, such as for infection or for post-operative complications
2. Severe Pulmonary Hypertension (PAH) (pulmonary pressure greater than 2/3 systemic) as defined by either echocardiogram (ECHO), or cardiac catheterizations or a CT-Angiogram consistent with PAH within the last 3 weeks.
3. Pneumothorax (active air leak) requiring chest tube within 72 hours of T=0
4. Active pulmonary hemorrhage within 72 hours of T=0
5. History of Grade III/IV interventricular hemorrhage without resolution or stability within 3 weeks of verifying eligibility
6. Severe congenital heart disease compromising pulmonary circulation
7. Other major congenital malformation (including but not limited to CDH) or known genetic syndromes at the discretion of the investigator
8. Use of an investigational drug within 7 days prior to confirmation of eligibility.
9. The clinical attending physician believes it is not in the subject's and/or parents/guardians best interest to participate in the trial.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Sustained oxygen desaturations for greater than ten minutes without response to increased oxygen therapy | Day 5, Day 10
  Incidence of sustained (greater than 10 minutes) oxygen desaturation events without response to increased oxygen therapy. These incidences will be measured by a continuous non-invasive percutaneous oxygen saturation monitor.
Persistent hypotension without response to volume expansion and/or inotropic therapy | Day 5, Day 10
  Incidence of persistent hypotension without response to volume expansion and/or inotropic therapy. Hypotension is a decrease in systolic blood pressure deemed significant by clinical staff. Measurement will be performed with a standard intensive care unit blood pressure cuff.
Change in number of major mucus plugging events | Day 5, Day 10
  Incidence of airway obstruction of the endotracheal tube, as indicated by decreased chest movement during mechanical ventilation, need for increased ventilator pressure, and/or elevation of carbon dioxide levels in the blood. Mucus plugs are confirmed by endotracheal suctioning.
Incidence of pneumothorax or pleural effusion with PFOB | Day 5, Day 10
  Incidence of pneumothorax in the child will be measured by transillumination of the chest and confirmed by chest x-ray.
Number of participants with sustained hypercapnia (elevated carbon dioxide in the blood, greater than 95 mmHg, for over four hours). | Day 5, Day 10
  Hypercapnia will be measured with blood tests and/or cutaneous carbon dioxide monitor.

SECONDARY OUTCOMES:
Change in fraction of inspired oxygen (FiO2) | Day 5, Day 10
  Fraction of inspired oxygen is the percentage of oxygen that the patient is receiving for his or her lung disease. An FiO2 of 0.21 is room air oxygen and 1.00 is 100% oxygen. The higher the FiO2, the more severe the respiratory disease.
Change in ventilator mean airway pressure (MAP) | Day 5, Day 10
  Mean airway pressure (MAP) is the average amount of airway pressure supplied to the lungs throughout a breath. Higher MAP indicates more severe disease.
Change in Respiratory Severity Score (MAP x FiO2) | Day 5, Day 10
  Respiratory Severity Score (RSS) is a scale computed as the Mean Airway Pressure (MAP) multiplied by the Fraction of Inspired Oxygen (FiO2). Clinically, the scale range will often lie between 1 and 10, with higher numbers indicating more severe disease. The RSS can theoretically reach a score as high as 30-35.

CONTACTS AND LOCATIONS:
Overall Officials: William Fox, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nocentini G, MacLaren G, Bartlett R, De Luca D, Perdichizzi S, Stoppa F, Marano M, Cecchetti C, Biasucci DG, Polito A, AlGhobaishi A, Guner Y, Gowda SH, Hirschl RB, Di Nardo M. Perfluorocarbons in Research and Clinical Practice: A Narrative Review. ASAIO J. 2023 Dec 1;69(12):1039-1048. doi: 10.1097/MAT.0000000000002017. Epub 2023 Aug 7. PMID 37549675